CLINICAL TRIAL: NCT05257772
Title: Electromechanically Optimised Right Ventricular Pacing In Hypertrophic Cardiomyopathy (EMORI-HCM)
Acronym: EMORI-HCM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 21HH7277
Record Dates: First submitted 2022-02-14; First posted 2022-02-25 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Hypertrophic Cardiomyopathy; Hypertrophic Obstructive Cardiomyopathy
Keywords: Right Ventricular Pacing; Atrio-Ventricular Delay; Dyssynchrony
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimum Right Ventricular Pacing On (Active Comparator): AV Delay Optimised RV Pacing. Subjects will remain in this arm for 3 months before being crossed-over.
  Interventions: Device: AV Delay Optimised RV Pacing
- Optimum Right Ventricular Pacing Off (No Intervention): Subjects will remain in this arm for 3 months before being crossed-over. The pacemaker will be programmed to minimum ventricular pacing & dynamic AV delay will be programmed off.

INTERVENTIONS:
Device: AV Delay Optimised RV Pacing — AV Delay Optimisation: will be performed using acute non-invasive blood pressure acquired using the Finometer device (Finapres Medical systems) and Echo to assess LVOT gradient change.
  Arms: Optimum Right Ventricular Pacing On

SUMMARY:
Hypertrophic Obstructive Cardiomyopathy (HOCM) is an inherited cardiac condition which causes the heart muscle to become abnormally thick causing obstruction of blood flow in the heart. This causes debilitating symptoms including shortness of breath, blackouts and chest pain. Current treatments are not ideal as the medication is often poorly tolerated or ineffective.

People with HOCM can often have an Implantable Cardioverter Defibrillator (ICD) to shock them out of dangerous arrhythmias. ICD's can also be used as pacemakers and are a promising treatment option, since they can alter the sequence of the heart muscle contraction thereby relieving the obstruction to the blood flow, making it easier for the heart to pump.

The study will recruit patients who already have an ICD/pacemaker or who are scheduled to have an ICD / pacemaker implanted. For patients who are due to have a device implanted high precision haemodynamic, echocardiographic and electrical measurement techniques will be used to assess whether adjusting the position of the pacing lead (at the time of implant) can bring about changes in LVOT gradient and blood pressure. These patients with a new device and also patients who already have a device in situ will then go on to have atrioventricular delay (AV Delay) optimisation so we can assess what the optimum AV delay should be programmed at in order to bring about the most improvement in LVOT gradient and blood pressure.

Patients will then be recruited into a medium term double blinded randomised crossover study. They will have optimum RV pacing settings turned on for 3 months. They will then return and be crossed over and have optimum RV pacing turned off for a further 3 months. The primary outcome will be to see if optimum RV pacing being turned on is effective in improving symptoms and quality of life.

DETAILED DESCRIPTION:
1. To test the impact of changing the pacing site and how it affects intra-ventricular delay and the amount of dyssynchrony.

   At the time of device implant, the RV lead will be positioned temporarily in the RV apex, low septum, high septum, RV free wall and coronary sinus. Non-invasive blood pressure will be measured by a Finometer device and Echo will assess LVOT gradient whilst pacing is turned on at each site. Ultra-high frequency ECG will be used to assess intraventricular dyssynchrony at each site. Haemodynamic measurements will also be made of aortic pressure and flow using a Combowire (with temporary heparinisation) to assess if non-invasively measured beat-by-beat finometer blood pressure are consistent with invasively measured changes in aortic flow. Combining these measurements will further assess the relationship between level of dyssynchrony, blood pressure and LVOT gradient change. The RV lead will then be implanted in a conventional position.
2. To use high-precision techniques to assess the impact of adjusting the AV Delay and how it affects blood pressure and LVOT gradient change.

   After patients have had their device implanted & those patients who already have a device in situ will then undergo an AV optimisation protocol (paced alternations of AV delay will be made from 40ms in 40ms increments up to 200ms / fusion). Non-invasive blood pressure will be measured (using a Finometer) along with LVOT gradient change with Echo at each AV delay and allow to identify the optimum AV Delay that brings about the most benefit in these acute parameters.
3. To follow patients over a period of 6 months in a double blinded randomised crossover trial. Patients will have active optimum RV pacing for 3 months. After this point they will then be crossed over for a further 3 months to optimum RV pacing off. Patient and assessor will remain blinded throughout. Patients will have the following assessed at baseline, 3 months and then at 6 months:

   * A symptom questionnaire (Kansas City Questionnaire + EQ5D5L Questionnaire). A smart phone symptom application will also record their daily symptoms during the 6 months follow up.
   * A blood test for BNP
   * A 6 Minute Walk Test & Cardiopulmonary Exercise test (MVOT)
   * An Echo scan
   * Device interrogation

Through simulation of a mixed-effects model to analyse the cross-over design, 60 patients would provide approximately 83% power.

ELIGIBILITY:
Inclusion criteria:

* All patients will have a clinical diagnosis of HOCM with an LVOT gradient of at least 30 mmHg, at rest or provoked.
* Symptomatic patients
* Can have co-existing mid-cavity obstruction.
* HOCM patients referred for Dual Chamber Pacemaker / ICD Implantation.
* Adults willing to take part (ages 18 - 100 years old)
* Able to give consent.

Exclusion criteria:

* Unable to give consent
* Children age < 18 years or adults > 100 years old
* Pregnant patient
* Patients with persistent Atrial Fibrillation or high grade Atrio-Ventricular Block

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-05-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
Patient symptoms | 6 months
  Patient symptoms via patient questionnaire - Kansas City Cardiomyopathy Questionnaire. All Kansas City Cardiomyopathy Questionnaire scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent

SECONDARY OUTCOMES:
Exercise Capacity | 6 months
  Change in exercise capacity by 6 Minute Walk Test
Exercise Capacity | 6 months
  Change in exercise capacity by Cardiopulmonary Exercise Testing (MVOT)
BNP | 6 months
  Change in BNP - Brain Natriuretic Peptide (blood test)
Patient preference of optimum pacing on or pacing off | 6 months
  An exploratory secondary outcome - patients will be asked at the end of the study which 3 month period they preferred (they will not be told during which 3 month period they were paced and not paced when they answer this question).
Patient symptoms | 6 months
  Patient symptoms via patient questionnaire - EQ-5D-5L Questionnaire. EQ-5D-5L health states can be summarised using the 5-digit code or represented by a single summary number (index value), which reflects how good or bad a health state is according to the preferences of the general population of a country/region. Most EQ-5D value sets have been obtained from a standardised valuation exercise, in which a representative sample of the general population in a country/region is asked to place a value on EQ-5D health states.
Patient symptoms | 6 months
  Patient symptoms via a smartphone daily symptom application
Echo Parameters | 6 months
  Change in LV Ejection Fraction (measured by Simpson's Biplane %)
Echo Parameters | 6 months
  Change in resting and peak exertion LVOT gradients (measured by Echo in mm Hg)
Pacemaker / ICD Activity Data | 6 months
  The pacemaker / device will be interrogated to give us information about participants activity levels (hrs per day)

CONTACTS AND LOCATIONS:
Overall Officials: Zachary I Whinnett, MRCP PhD, Principal Investigator — Imperial College London
Locations (1):
- National Heart & Lung Institute, Imperial College London, London, United Kingdom

REFERENCES:
- [Background] Arnold AD, Howard JP, Chiew K, Kerrigan WJ, de Vere F, Johns HT, Churlilov L, Ahmad Y, Keene D, Shun-Shin MJ, Cole GD, Kanagaratnam P, Sohaib SMA, Varnava A, Francis DP, Whinnett ZI. Right ventricular pacing for hypertrophic obstructive cardiomyopathy: meta-analysis and meta-regression of clinical trials. Eur Heart J Qual Care Clin Outcomes. 2019 Oct 1;5(4):321-333. doi: 10.1093/ehjqcco/qcz006. PMID 30715300
- [Background] Slade AK, Sadoul N, Shapiro L, Chojnowska L, Simon JP, Saumarez RC, Dodinot B, Camm AJ, McKenna WJ, Aliot E. DDD pacing in hypertrophic cardiomyopathy: a multicentre clinical experience. Heart. 1996 Jan;75(1):44-9. doi: 10.1136/hrt.75.1.44. PMID 8624871
- [Background] Breithardt G. MADIT-CRT (Multicenter Automatic Defibrillator Implantation Trial-Cardiac Resynchronization Therapy): cardiac resynchronization therapy towards early management of heart failure. Eur Heart J. 2009 Nov;30(21):2551-3. doi: 10.1093/eurheartj/ehp383. Epub 2009 Sep 22. No abstract available. PMID 19773224
- [Background] Kyriacou A, Pabari PA, Whinnett ZI, Arri S, Willson K, Baruah R, Stegemann B, Mayet J, Kanagaratnam P, Hughes AD, Francis DP. Fully automatable, reproducible, noninvasive simple plethysmographic optimization: proof of concept and potential for implantability. Pacing Clin Electrophysiol. 2012 Aug;35(8):948-60. doi: 10.1111/j.1540-8159.2012.03435.x. Epub 2012 Jul 2. PMID 22747698
- [Background] Jurak P, Curila K, Leinveber P, Prinzen FW, Viscor I, Plesinger F, Smisek R, Prochazkova R, Osmancik P, Halamek J, Matejkova M, Lipoldova J, Novak M, Panovsky R, Andrla P, Vondra V, Stros P, Vesela J, Herman D. Novel ultra-high-frequency electrocardiogram tool for the description of the ventricular depolarization pattern before and during cardiac resynchronization. J Cardiovasc Electrophysiol. 2020 Jan;31(1):300-307. doi: 10.1111/jce.14299. Epub 2019 Dec 5. PMID 31788894
- [Background] Whinnett ZI, Francis DP, Denis A, Willson K, Pascale P, van Geldorp I, De Guillebon M, Ploux S, Ellenbogen K, Haissaguerre M, Ritter P, Bordachar P. Comparison of different invasive hemodynamic methods for AV delay optimization in patients with cardiac resynchronization therapy: implications for clinical trial design and clinical practice. Int J Cardiol. 2013 Oct 3;168(3):2228-37. doi: 10.1016/j.ijcard.2013.01.216. Epub 2013 Mar 5. PMID 23481908
- [Derived] Mohal JS, Whinnett ZI, Mohiddin SA, Malcolmson J, Elliott P, Ormerod JOM, Prasad S, Ware JS, Cooper RM, Tanner MA, Khalique Z, Shah JS, Keene D, Tangkongpanich P, Lewis EC, Sharma C, Reddy RK, Naraen A, Saleh K, Samways JW, Howard JP, Artico J, Kanagaratnam P, Francis DP, Al-Lamee RK, Varnava A, Shun-Shin MJ, Arnold AD. Electromechanically Optimized Right Ventricular Pacing for Obstructive Hypertrophic Cardiomyopathy: The EMORI-HCM Trial. J Am Coll Cardiol. 2026 Jan 20;87(2):124-139. doi: 10.1016/j.jacc.2025.08.050. Epub 2025 Aug 31. PMID 40892619